CLINICAL TRIAL: NCT00414622
Title: A Double Blind, Placebo-Controlled Randomized Study to Compare the Safety and Tolerability of GTS-21 (25 Mg TID, 50 Mg TID, 75 Mg TID and 150 Mg TID) When Administered Daily for 28 Days to Participants With Probable Alzheimer's Disease
Brief Title: GTS21-201 for Alzheimer Disease:GTS-21 Administered Daily for 28 Days to Participants With Probable Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CoMentis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GTS21-201
Expanded Access: Available
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2006-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; Probable Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 3-(2,4-dimethoxybenzylidene)anabaseine

INTERVENTIONS:
Drug: DMXB-A

SUMMARY:
A Double Blind, Placebo-Controlled Randomized Study to Compare the Safety and Tolerability of GTS-21 (25 Mg TID, 50 Mg TID, 75 Mg TID and 150 Mg TID) When Administered Daily for 28 Days to Participants With Probable Alzheimer's Disease

DETAILED DESCRIPTION:
A Double Blind, Placebo-Controlled Randomized Study to Compare the Safety and Tolerability of GTS-21 (25 Mg TID, 50 Mg TID, 75 Mg TID and 150 Mg TID) When Administered Daily for 28 Days to Participants With Probable Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

* probable Alzheimer

Exclusion Criteria:

* others

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
CDR

SECONDARY OUTCOMES:
ADAS-cog

CONTACTS AND LOCATIONS:
Overall Officials: Henry Hsu, MD, Study Director — CoMentis
Locations (1):
- Clinical Dept., 280 South San Francisco, California, United States